CLINICAL TRIAL: NCT02875210
Title: Comparative Study of Anterior Tibial Translation Measurement by Four Different Laximeters in Anterior Cruciate Ligament Ruptures
Brief Title: Comparative Study of Anterior Tibial Translation Measurement by Four Laximeters in Anterior Cruciate Ligament Ruptures
Acronym: LAXIMETRIE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Versailles Hospital (Other)
Responsible Party: Principal Investigator, Nicolas Pujol, Investigator coordinator, Versailles Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P15/02_LAXIMETRIE
Record Dates: First submitted 2016-08-11; First posted 2016-08-23 (Estimated); Last update posted 2016-08-23 (Estimated); Status verified 2016-08

CONDITIONS: Anterior Cruciate Ligament Rupture
Keywords: Anterior Cruciate Ligament; A02.835.583.512.100
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patient with anterior cruciate ligament rupture (Experimental): Anterior laxity of patient was measure with 4 laximeters:Telos, reference laximeter and with three other instruments called, KT-1000, GnrB and Rolimeter.
  Interventions: Procedure: Laximeter measurement

INTERVENTIONS:
Procedure: Laximeter measurement

SUMMARY:
Actually, there are several laximeters for measuring anterior tibial translational in case of anterior cruciate ligament rupture. The most commonly used are telos, KT-1000, GnrB and Rolimeter. Results of these instrumented tests, which expressed in differential (millimeters values), have a bad correlation between them and so are not comparable in current literature. The aim of this study was to compare results of these tests and establish a ratio (pathologic knee laxity/ healthy knee laxity) to reduce differences between each instrumented test.

ELIGIBILITY:
Inclusion Criteria:

* Obtaining a written informed consent of the patient,
* Affiliated with a Medicare (or rightful beneficiary),
* Disponibility of the patient,
* Patients ≥ 18 ans,
* Anterior cruciate ligament rupture concerned only one knee of the patient.

Exclusion Criteria:

* Patient is in the exclusion period for another study,
* Patient is under judicial protection, guardianship, or curators,
* Eligible patients who are refused to sign consent,
* It is impossible to give clear informations to the patient,
* Pregnant women,
* Nursing mother,
* Patient which has been already operate of the other knee,
* Patient present ligament lesions associated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2015-07; Primary Completion 2017-01 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Comparison of anterior laxity measurement between pathologic and healthy knees. | 18 months
  Collect and compare differential values of anterior laxity between pathologic and healthy knee obtained by four different laximeters (Telos, KT-1000, GnrB and Rolimeter)

SECONDARY OUTCOMES:
Sensivity and specificity of each instrument | 18 months
  Determine sensivity and specificity of each instrument test to highlight a cruciate ligament rupture and find the better test.
  Evaluations are using the 4 following devices: Telos ©, KT-1000 ©, Rolimeter, and GnrB.
Correlation between the f4 laximeters results | 18 months
  Estimate if correlation between two results increase discriminating capacity in comparison with the reference.
Value of the ratio : pathologic (anterior knee laxity) versus healthy knee | 18 months
  Compare ratio pathologic versus healthy knee obtained with each instrument to determine a possible harmonization of measurements

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas PUJOL, MD, Principal Investigator — Central Hospital of Versailles
Locations (1):
- Centre Hospitalier de Versailles, Le Chesnay, France

IPD SHARING:
Plan to Share IPD: Undecided